CLINICAL TRIAL: NCT02436551
Title: Gestational Diabetes in Central Asia: Prevalence and Management
Acronym: GESDICA
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Helmholtz Zentrum München (Industry)
Responsible Party: Principal Investigator, Klaus Parhofer, Professor of Endocrinology and Metabolism, Ludwig-Maximilians - University of Munich
Other Study IDs: GESDICA
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women in Tajikistan
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
Evaluate prevalence and management of gestational diabetes in Tajikistan in two different settings (one rural and one urban).

ELIGIBILITY:
Inclusion Criteria:

* pregnancy

Exclusion Criteria:

* known diabetes mellitus

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women in rural setting; pregnant women in urban setting;
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
prevalence of gestational diabetes | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Med. Dept. 2, University Munich, Munich, Germany